CLINICAL TRIAL: NCT00588042
Title: Remote Myocardial Ischemic Preconditioning in Humans
Acronym: RemoteMIPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Abhiram Prasad, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-005081
Record Dates: First submitted 2007-12-21; First posted 2008-01-08 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Ischemia
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; Coronary Artery Disease; Coronary Occlusion
MeSH Terms: conditions — Coronary Artery Disease; Coronary Occlusion | interventions — Sphygmomanometers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Arm ischemia will be induced using a blood pressure cuff that will be placed around the upper part of the arm, and inflated to 200 mm Hg for 3-minutes and then deflated for 3-minutes
  Interventions: Device: Blood pressure cuff
- 2 (Sham Comparator): 3-cycles of cuff inflation (10 mmHg)-deflation will also be performed in the control group for similar durations without inducing ischemia
  Interventions: Device: blood pressure cuff

INTERVENTIONS:
Device: Blood pressure cuff — Arm ischemia will be induced using a blood pressure cuff that will be placed around the upper part of the arm, and inflated to 200 mm Hg for 3-minutes and then deflated for 3-minutes
  Other Names: sphygmomanometer
  Arms: 1
Device: blood pressure cuff — 3-cycles of cuff inflation (10 mmHg)-deflation will also be performed in the control group for similar durations without inducing ischemia
  Other Names: sphygmomanometer
  Arms: 2

SUMMARY:
Ischemic preconditioning (IP) has been shown in animal studies to increase the myocardial tolerance to subsequent ischemia. Our primary hypothesis is that remote IP reduces myocardial ischemic injury during PCI.

DETAILED DESCRIPTION:
Our primary hypothesis is that remote IP reduces myocardial ischemic injury during PCI. We will also test the hypotheses that IP diminishes the inflammatory response to PCI, and that higher baseline blood endothelial progenitor cell counts are predictive of a favorable response to IP.

Aim 1: To evaluate whether remote ischemic preconditioning reduces the frequency of myonecrosis (troponin T≥0.03 ng/ml following PCI).

Aim 2: To evaluate whether remote ischemic preconditioning reduces the inflammatory response to PCI (post PCI hsCRP level).

Aim 3: To evaluate whether pre-procedure circulating endothelial progenitor cell counts correlate with the effect of remote ischemic preconditioning on myonecrosis.

Background: Percutaneous coronary intervention (PCI) frequently results in ischemic myonecrosis. Ischemic preconditioning (IP) has been shown in animal studies to increase the myocardial tolerance to subsequent ischemia. Our primary hypothesis is that remote IP reduces myocardial ischemic injury during PCI.

Aims: The aims of the study are to assess in patients with coronary artery disease requiring PCI, whether remote IP reduces: 1) the frequency of myonecrosis; and 2) the inflammatory response to PCI; and 3) whether the effect of IP correlates with pre-procedure circulating endothelial progenitor cell counts.

Methods: The study is a prospective, randomized trial to assess the efficacy of remote IP as adjunctive non-pharmacological therapy for PCI in patients with stable or unstable angina. Remote IP will be performed by 3 cycles of 3-minutes of arm ischemia alternating with 3- minutes of reperfusion of the arm immediately before PCI. Myonecrosis and inflammation will be detected by measuring serum troponin T and high sensitivity C-reactive protein, respectively. Blood EPC counts will also be measured before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for randomization if they meet the following criteria:

  1. Age ≥ 18 years
  2. Clinically indicated elective or urgent PCI

Exclusion Criteria:

* Patients will be ineligible for the study if one or more of the following conditions exist:

  1. Pre-PCI Troponin T ≥ 0.03
  2. Systemic hypotension (systolic <90 mmHg) or cardiogenic shock
  3. Presence of an arteriovenous fistula or lymphedema of either arm
  4. Currently enrolled in other active cardiovascular investigational studies
  5. Severe endocrine, hepatic, renal, disorders
  6. Pregnancy or lactation
  7. Inability to provide consent
  8. Federal Medical Center inmates
  9. Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Post PCI myonecrosis measured as a maximum troponin T ≥0.03 | 16 hours post PCI

SECONDARY OUTCOMES:
Post PCI myonecrosis measured as an elevation in creatine kinase MB fraction (CK-MB> 1 X upper limit of normal) | 16 hours post procedure
Magnitude of ST segment elevation on an intracoronary electrocardiogram during balloon inflation | During PCI procedure
Coronary perfusion measured as coronary flow reserve derived from TIMI frame counts | During PCI
Blood high sensitivity C-reactive protein level | Immediately prePCI
Blood endothelial progenitor cell counts (EPC) | Immediately prePCI

CONTACTS AND LOCATIONS:
Overall Officials: Abhiram Prasad, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Prasad A, Gossl M, Hoyt J, Lennon RJ, Polk L, Simari R, Holmes DR Jr, Rihal CS, Lerman A. Remote ischemic preconditioning immediately before percutaneous coronary intervention does not impact myocardial necrosis, inflammatory response, and circulating endothelial progenitor cell counts: a single center randomized sham controlled trial. Catheter Cardiovasc Interv. 2013 May;81(6):930-6. doi: 10.1002/ccd.24443. Epub 2012 Nov 8. PMID 22517646